CLINICAL TRIAL: NCT07036848
Title: The Efficacy and Safety of Surgical Treatment in Type IVa Congenital Biliary Dilation: A Multi-center Cohort Study
Brief Title: Efficacy and Safety of Surgical Treatment for Type IVa CBD
Status: Recruiting | Type: Observational
Sponsor: Beijing Tsinghua Chang Gung Hospital (Other)
Responsible Party: Principal Investigator, Shuo Jin, Associate Chief Physician, Beijing Tsinghua Chang Gung Hospital
Other Study IDs: 24637-0-01
Record Dates: First submitted 2025-06-17; First posted 2025-06-25 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Choledochal Cyst
Keywords: Biliary Dilatation, Cohort Study, Surgical Treatment
MeSH Terms: conditions — Choledochal Cyst

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Liver Resection Group: This group included patients with type IVa BD who underwent liver resection, extrahepatic bile duct resection and Roux-en-Y hepaticojejunostomy
- Hepaticojejunostomy Group: This group included patients with type IVa BD who underwent extrahepatic bile duct resection and Roux-en-Y hepaticojejunostomy

SUMMARY:
This study is a multicenter, bidirectional cohort study aimed at continuously enrolling patients with biliary dilatation from 25 medical centers in China. It will collect comprehensive life-cycle data from the cohort to establish a Chinese cohort for IVa biliary dilatation (BD). Based on this cohort, the study seeks to compare the perioperative risks, long-term outcomes, and quality of life of type IVa BD following surgical treatment, to establish standardized surgical treatment strategies for type IVa BD.

DETAILED DESCRIPTION:
Biliary dilatation (BD) is a common complex benign biliary disease. The incidence rate in Asia is one of every 1000 individuals, and the incidence rate in Europe and America is about one of every 50,000-150,000 individuals. Type IVa BD was the most commonly intrahepatic BD and the second most commonly identifiable cyst type. According to the Todani classification of congenital type IVa represents a combination of intra-and extrahepatic cystic ectasias.

However, there is still significant controversy regarding the surgical treatment approaches for this disease. Current treatment methods mainly include hepaticojejunostomy and hepatectomy. On the one hand, studies suggest that performing hepaticojejunostomy while relieving hilar bile duct stricture is sufficient. Previous research has reported that intrahepatic bile duct cysts may regress after hepaticojejunostomy. However, recent studies have described that type IV-A bile duct (BD) patients may develop long-term complications such as intrahepatic bile duct stones, anastomotic stricture, and cholangitis after hepatojejunostomy, although the specific incidence rates remain unclear. On the other hand, only a few small-series studies have reported that hepatectomy may achieve satisfactory efficacy in treating intrahepatic BD. Nevertheless, other studies have shown that 30% of patients may develop postoperative intrahepatic bile duct stones. Considering that this procedure is a higher-risk surgery compared to bilioenteric anastomosis, its effectiveness and safety in the treatment of type IVa BD introduce greater uncertainty.

This study aims at enrolling patients with biliary dilatation from 25 medical centers in China. It will collect comprehensive life-cycle data from the cohort to establish a Chinese cohort for IVa BDs. Based on this cohort, the study seeks to compare the perioperative risks, long-term outcomes, and quality of life of type IVa BD following surgical treatment, to establish standardized surgical treatment strategies for type IVa BD.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have been diagnosed with Todani type IVa BD.
2. Patients aged between 0 and 80 years old, regardless of gender.
3. First-time receipt of surgery.

Exclusion Criteria:

1. With abnormal intrapancreatic bile duct
2. Inappropriate Roux-loop length (outside the range of 40-60 cm for adults and 15-30 cm for children)
3. With non-relevant surgical interventions
4. Pathologically confirmed carcinogenesis
5. Unresolved choledocholithiasis, bile duct stenosis, and Intrahepatic bile duct stones during the procedure.
6. Unavailable follow-up information.

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with a definitive diagnosis of Todani type IVa biliary dilation in the participating centers
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2025-07-14 (Actual); Primary Completion 2025-07-14 (Actual); Study Completion 2035-07-01 (Estimated)

PRIMARY OUTCOMES:
Long-term complication-free survival (LCFS) | After 30 or 90 days of surgery
  For patients who have undergone surgical treatment, the occurrences of long-term postoperative complications include recurrent cholangitis, intrahepatic bile duct stones, stenosis of the bilioenteric anastomosis, and other such conditions

SECONDARY OUTCOMES:
Overall perioperative complication rate | Within 30 or 90 days postoperatively
  The occurrence of perioperative complications, including bile leakage, pancreatic leakage, liver failure, bacteremia, abdominal fluid accumulation, and intra-abdominal infections, among others
Malignant transformation rate | Through study completion, an average of 1 year
  The occurrence of malignant transformation associated with bile duct dilatation
Mayo Score | Through study completion, an average of 6 months
  Long-term outcome was evaluated according to the dedicated clinical evaluation score reported by the Mayo Clinic: excellent, if the patient remained free of symptoms without further reintervention; good, if the patient had occasional and mild episodes of cholangitis or pancreatitis, which were not impairing the quality of life; fair, if the patient had repeated episodes of cholangitis or pancreatitis,or portal hypertension without further reintervention; poor, if the patient required later biliary or liver-related surgical procedures, developed biliary cirrhosis or complications because of portal hypertension, or died from cyst-related malignancy or liver and biliary-related complications.
Severe perioperative complication rate | Within 30 or 90 days postoperatively
  The occurrence of severe perioperative complications (Clavien-Dindo grading ≥ III), including bile leakage, pancreatic leakage, liver failure, bacteremia, abdominal fluid accumulation, and intra-abdominal infections, among others.
Reoperation rate | After 30 or 90 days of surgery
  The occurrence of reoperation after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Shuo Jin, PhD, Principal Investigator — Beijing Tsinghua Changgeng Hospital
Locations (1):
- Beijing Tsinghua Changgung Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No